CLINICAL TRIAL: NCT03901612
Title: Evaluation of a Peri-Operative Continuous Bilateral Erector Spinae Plane (ESP) Continuous Catheter After Open Cardiac Surgery in Adults
Brief Title: Erector Spinae Catheter for Open Heart Surgery
Acronym: ESPADULT2
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: covid and surgeon left
Sponsor: Vinmec Healthcare System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VINMECCP
Record Dates: First submitted 2019-04-02; First posted 2019-04-03 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Post Operative Analgesia

STUDY DESIGN:
Intervention Model Description: Randomized Controlled double blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Solution infused prepared by a different team with a rescue envelop to open in case of incident
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saline solution (Placebo Comparator): Post operative analgesia throw the thoracic Erector spinae catheter with saline solution and opioid rescue
  Interventions: Drug: saline 09%
- Ropivacaine (Experimental): Post operative analgesia throw the thoracic Erector spinae catheter with Ropivacaine 0.2% solution and opioid rescue
  Interventions: Drug: Ropivacaine 0.2%

INTERVENTIONS:
Drug: Ropivacaine 0.2% — Continuous post operative regional analgesia
  Arms: Ropivacaine
Drug: saline 09% — Continuous post operative regional analgesia
  Arms: Saline solution

SUMMARY:
Fast track to Extubation after cardiothoracic surgery is becoming more common after a number of reports showing it is safe and effective. However, It has introduced new challenges to pain control. Intubated patients require larger doses of opioids and benzodiazepines for comfort. In patients who are awake and spontaneously breathing, pain and agitation cannot be treated with lower doses.

Some centers still administer continuous infusions of opioid and benzodiazepines to extubated patients. These infusions may not be necessary and may even be harmful.

The recent pilot study (In press in Journal of cardio thoracic vascular anesthesia ) in our Vinmec hospitals performing open heart surgeries of peri-operative regional analgesia by Continuous Bilateral Erector Spinae Plane Blocks in adult showed that the pain relief was efficient and the requirement for opioids was zero in post-operative period.

It confirmed that the impact of regional anesthesia techniques on main procedure-specific postoperative outcomes is very important in opioids decreased use in the context of fast-track programs that are fully suggested after cardiac surgery.

In April 2017 we introduced the technique of ESP block for open heart surgeries in Adults and in pediatric. At the beginning we performed single shot block and the patients still needed during around 30 to 40 hours small doses of opioids to release their pain according to the evaluation by Comfort-B,FLACC VAS Scales. Since we are performing continuous peri-operative regional analgesia by Bilateral ESP catheters the requirement for additional opioids to release the pain is zero based on our practice of 480 ESP catheters for open heart surgeries.

We would like to compare the 2 analgesic techniques and analyze the post operative opioid consumption, the quality of recovery and the quality of life after the surgery.

DETAILED DESCRIPTION:
Methodology With the Approval of Ethical committee of VinMec Healthcare and after Patient's information and consent from guardian or parents, adults will be randomized via a random number generator into one of two treatment groups by the person who obtained consent which is prescribed in the nurse preparation file".

Group 1: will receive a single shot dose of local anesthetic Ropivacaine throw ESP catheters and 6 hours after continuous infusion of Iso saline with a rescue analgesia in case of pain according to the bellow protocol Group 2 :will received a single shot dose of local anesthetic Ropivacaine throw ESP catheters and 6 hours after a continuous infusion of Ropivacaine with a rescue analgesia if needed according to the bellow protocol Catheter Performance The anesthesia team will perform to all patients without exclusion criteria (Group I & II) for open heart surgery after the anesthesia induction a bilateral insertion of an Erector Spinae Plane Block catheter under ultrasound guidance.

Patient in right lateral decubitus. The anesthesiologist will use an Ultrasound linear probe at T4 level and identify the T4 transverse process. By hydro-dissection he will identify the inter-fascial space between the Inter-transverse ligament anteriorly and the Erector Spinae Muscle posteriorly to insert under ultrasound vision a catheter . The tip of the catheter should be at T5 Transverse level seen by ultrasound. The anesthesiologist check the right position of the catheter with a dextrose 5% injection = 1 to 3 mL under ultrasound vision and see the spread of the dextrose in the inter-fascial space which sign that the catheter is not intra-vascular. This procedure will be bilateral. The catheter will have a yellow label on the Huer®-Lock connector to identify clearly that it is regional analgesia catheter to prevent any errors of miss injection. (Yellow is the international identification of regional anesthesia analgesia lines).

After this control an induction low dose is injected. Table 1 Induction dose Patient 30 - 40 kg = 6 mL of Ropivacaine 0.5% / side Patient 40 - 50 kg = 8 mL of Ropivacaine 0.5% / side Patient 50 - 60 kg = 10 mL of Ropivacaine 0.5% / side Patient 60 - 70 kg = 12 mL of Ropivacaine 0.5% / side Patient > 70 kg = 14 mL of Ropivacaine 0.5% / side 5h after, the ESP catheter induction, prepare the solution in the pump The clinical research nurse specially trained for this study will proceed to the randomization of the patient according to the randomization table and prepare the solution in the pump as per attached protocol. They will put the number of patient's randomization on the pump. The nurse receives instruction to keep strictly confidential the content of the pumps. They will deliver the prepared pumps to the anesthesiologist and anesthesia nurse in charge of the patient. They will connect the pumps to the patient and start the infusion 6 hours after as per protocol.

Group 1 & Group 2 will have the blinded solution in the pump ♣ Table 2 Intermittent Automatic bolus For post operative ESP catheter infusion Patient 30 - 40 kg = 6 mL of Ropivacaine 0.5% / side/ 6h Patient 40 - 50 kg = 8 mL of Ropivacaine 0.5% / side/ 6h Patient 50 - 60 kg = 10 mL of Ropivacaine 0.5% / side/ 6h Patient 60 - 70 kg = 12 mL of Ropivacaine 0.5% / side/ 6h Patient > 70 kg = 14 mL of Ropivacaine 0.5% / side/ 6h (The bolus on the second catheter will be delayed by 1 hour).

* Assess Pain Level All the participants to this studies were trained to the protocol last January 2018 and the nurse trained to random performance and data collection. For all groups . The nurse will assess pain level at rest and mob after extubation and also the Localization of the pain

  * Sternum
  * Back pain
  * Drains If pain FLACC > 3 or VAS at rest or at Mob >4

    * If Extension problem increase IAB 2 mL/catheter of the solution inside the pump (DOUBLE BLINDED neither the patient, the physician in charge of the patient and the investigator know what is in the pump .on the side concerned (by increasing the volume we will increase the extension of the analgesia block. This volume increasing will be limited to only one increase. If still pain after the anesthesiologist is not allowed to increase again the volume and should shift to rescue analgesia described below)
    * IF Not the patient will receive a dose of morphine as follow :

Morphin 50 mcg/kg/min if patient is still intubated

Morphine PCA mode rescue : if patient extubation:

* Concentration : 50 mg/50 ml
* Loading dose: 1mg
* PCA dose demand: 1 mg/dose
* Lockout: 10 min
* Continuous rate (basal): 0 Dose limit (hr): 6mg/hour Pain Re-assessment 1 hour after settings changes of the pump

  * if the FLACC < 3 or VAS inferior to 4 : continue ESP catheters and paracetamol+ ibuprofen /6h
  * if the FLACC >3 VAS > 4= poor analgesia +> Rescue analgesia by opioids as before this technique and commonly used in open heart surgeries. Morphine 30 mcg/kg/h.
* Catheter Removal A Bi-daily inspection of the catheters insertion points will be done. If redness around puncture point the catheters will be removed and shift to classical IV analgesia to prevent any infection. It will be declared as a minor incident in the study.

ESP catheters will be removed 2 hours after drain removal maximum 56h after insertion.

2 h. after Drain removal and ESP catheter removed the analgesia in both group will be with the following antalgics:

* Paracetamol Systematically 1g/6h
* Ketorolac 30 mg IV every 8h ♣ Scales evaluate the pain:

  * Before extubation FLACC scale at rest
  * After extubation and still drains will remain we will use VAS Scale at rest and at Mob (sitting in bed rotation of the thorax) Localization of the pain
* Sternum
* Back pain
* Drains ¬ After drains removal we will use FLACC Scale rest and Mob ( sitting in bed rotation of the thorax) and pain localization A check list anesthesia protocol will be provided for each patient and check list for the pump solution will be provided for the nurse in charge of randomization and preparation of the pump ♣ Statistical analysis and sample size calculation Based on our prior institutional unpublished retrospective data of maximal pain scores from 24 - 48 hours post-surgery in patients who received Single shot ESP bl0cks who underwent open heart surgeries (mean 3 with standard deviation 2.2) We determine that a total of 18 patients per arm will be needed to achieve A decrease in mean pain of 1.5 with 80% power with 5% alpha. We will assume up to 10% lost to follow up and 10% of patients would be non-compliant so we will enroll 25 patients in each group.

ELIGIBILITY:
Inclusion Criteria:

* all patients having an elective open heart surgery

Exclusion Criteria:

* refusal of the patient allergy to local anesthetics instable patient

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-05 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | From extubation to 48 hours after end of surgery
  Morphine consumption in milligrams

SECONDARY OUTCOMES:
Quality of recovery after the surgery | 48 hours after end of surgery
  Quality of post operative recovery using the table QOR15* from 0 to 15
Quality of Life after the surgery | 30 days after end of surgery
  Quality of post operative life using the table QOL36* from 0 to 36
post operative pain | every 6 hours during 48hours after the end of the surgery
  Level of pain at rest and at mobilization using Visual analogic scale

CONTACTS AND LOCATIONS:
Overall Officials: sebastien bertin, md, Study Chair — VinMec HS
Locations (1):
- VinMec INternational hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alghamdi AA, Singh SK, Hamilton BC, Yadava M, Holtby H, Van Arsdell GS, Al-Radi OO. Early extubation after pediatric cardiac surgery: systematic review, meta-analysis, and evidence-based recommendations. J Card Surg. 2010 Sep;25(5):586-95. doi: 10.1111/j.1540-8191.2010.01088.x. PMID 20626510
- [Background] Garg R, Rao S, John C, Reddy C, Hegde R, Murthy K, Prakash PV. Extubation in the operating room after cardiac surgery in children: a prospective observational study with multidisciplinary coordinated approach. J Cardiothorac Vasc Anesth. 2014 Jun;28(3):479-87. doi: 10.1053/j.jvca.2014.01.003. Epub 2014 Apr 18. PMID 24746595
- [Background] Heinle JS, Diaz LK, Fox LS. Early extubation after cardiac operations in neonates and young infants. J Thorac Cardiovasc Surg. 1997 Sep;114(3):413-8. doi: 10.1016/S0022-5223(97)70187-9. PMID 9305193
- [Background] Kin N, Weismann C, Srivastava S, Chakravarti S, Bodian C, Hossain S, Krol M, Hollinger I, Nguyen K, Mittnacht AJ. Factors affecting the decision to defer endotracheal extubation after surgery for congenital heart disease: a prospective observational study. Anesth Analg. 2011 Aug;113(2):329-35. doi: 10.1213/ANE.0b013e31821cd236. Epub 2011 Apr 13. PMID 21490084
- [Background] Carli F, Kehlet H, Baldini G, Steel A, McRae K, Slinger P, Hemmerling T, Salinas F, Neal JM. Evidence basis for regional anesthesia in multidisciplinary fast-track surgical care pathways. Reg Anesth Pain Med. 2011 Jan-Feb;36(1):63-72. doi: 10.1097/AAP.0b013e31820307f7. PMID 22002193
- [Background] Macaire P, Ho N, Nguyen T, Nguyen B, Vu V, Quach C, Roques V, Capdevila X. Ultrasound-Guided Continuous Thoracic Erector Spinae Plane Block Within an Enhanced Recovery Program Is Associated with Decreased Opioid Consumption and Improved Patient Postoperative Rehabilitation After Open Cardiac Surgery-A Patient-Matched, Controlled Before-and-After Study. J Cardiothorac Vasc Anesth. 2019 Jun;33(6):1659-1667. doi: 10.1053/j.jvca.2018.11.021. Epub 2018 Nov 19. PMID 30665850
- [Background] Tsui BCH, Navaratnam M, Boltz G, Maeda K, Caruso TJ. Bilateral automatized intermittent bolus erector spinae plane analgesic blocks for sternotomy in a cardiac patient who underwent cardiopulmonary bypass: A new era of Cardiac Regional Anesthesia. J Clin Anesth. 2018 Aug;48:9-10. doi: 10.1016/j.jclinane.2018.04.005. Epub 2018 May 26. No abstract available. PMID 29684728
- [Background] Biswas A, Luginbuehl I, Szabo E, Caldeira-Kulbakas M, Crawford MW, Everett T. Use of Serratus Plane Block for Repair of Coarctation of Aorta: A Report of 3 Cases. Reg Anesth Pain Med. 2018 Aug;43(6):641-643. doi: 10.1097/AAP.0000000000000801. PMID 29794944